Date: 2025-08-31

**Unique Protocol ID: 2024-07566-01** 

Title: The Time Before the Crime - Risk Patterns in Offenders Undergoing a Forensic

Psychiatric Evaluation (Tibec)

Principal Investigator: Katarina Howner, Associate professor, Karolinska Institutet

## **Statistical Analysis Plan**

To test the hypothesis regarding risk patterns, we will use a combination of tailored statistical tests, adjusting for potential confounders. Firstly, we will first calculate frequency distributions, means, and standard deviations for baseline characteristics. To compare variables between the groups, we will employ the chi-square test for categorical variables and t-test for numerical variables. The primary analysis will focus on assessing associations between specific risk factors and the likelihood of undergoing an FPE. Logistic regression will be central to this analysis. Furthermore, we will apply conditional logistic regression, a statistical method well-suited for matched case-control designs. By using conditional logistic regression, we will obtain precise odds ratios that quantify the strength of the association between risk factors and the likelihood of undergoing an FPE. Finally, to address the issue of potential missing data (e.g., incomplete psychiatric records), sensitivity analyses will be conducted, which will help determine how missing data might impact on the robustness and validity of the results.